CLINICAL TRIAL: NCT01069302
Title: Clopidogrel High Dose Evaluation for the Patient With Coronary Artery Disease in Japan
Acronym: CHOICE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeshi Morimoto (Other)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Professor, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: C369
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High loading and high maintenance (Active Comparator): Clopidogrel loading 600mg and maintenance 150mg for 7days
  Interventions: Drug: Clopidogrel
- High loading and low maintenance (Active Comparator): Clopidogrel loading 600mg and maintenance 75mg for 7days
  Interventions: Drug: Clopidogrel
- Low loading and high maintenance (Active Comparator): Clopidogrel loading 300mg and maintenance 150mg for 7days
  Interventions: Drug: Clopidogrel
- Low loading and low maintenance (Active Comparator): Clopidogrel loading 300mg and maintenance 75mg for 7days
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel loading 600mg and maintenance 150mg for 7days
  Arms: High loading and high maintenance
Drug: Clopidogrel — Clopidogrel loading 600mg and maintenance 75mg for 7days
  Arms: High loading and low maintenance
Drug: Clopidogrel — Clopidogrel loading 300mg and maintenance 150mg for 7days
  Arms: Low loading and high maintenance
Drug: Clopidogrel — Clopidogrel loading 300mg and maintenance 75mg for 7days
  Arms: Low loading and low maintenance

SUMMARY:
The purpose of this study is to evaluate the effect of high dose clopidogrel as the antiplatelet therapy on inhibition of platelet aggregation in Japanese patients scheduled for percutaneous coronary intervention due to ischemic heart disease.

DETAILED DESCRIPTION:
Dual antiplatelet therapy of aspirin and thienopyridine is used to prevent stent thrombosis after percutaneous coronary intervention (PCI). Clopidogrel is the most popular thienopyridine. Following the 300mg clopidogrel loading dose (LD) at first day, patients take 75mg maintenance dose (MD) to inhibit platelet aggregation after coronary stent implantation. 600mg high LD inhibit platelet aggregation more rapidly and strongly than standard LD and prevent thrombotic event around the PCI. Similarly high MD inhibit platelet aggregation more strongly. Interindividual variability of clopidogrel anti-platelet effect has been reported. In Japanese, there are many non or hyporesponders to clopidogrel compared to the Western population. The purpose of this study is to evaluate the effect of high dose clopidogrel as the antiplatelet therapy on inhibition of platelet aggregation in Japanese patients scheduled for PCI due to ischemic heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for percutaneous coronary intervention due to ischemic heart disease
* Patients taking aspirin 81-100mg at least 1 week.

Exclusion Criteria:

* Patients with ST elevation myocardial infarction
* Patients have contraindication of aspirin or clopidogrel
* Patients taking warfarin
* Patients received thrombolytic therapy within 2 weeks
* Patients taking anti-platelet agents except aspirin within 1 month
* Patients taking corticosteroid.
* Patients taking proton pump inhibitor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Inhibition of platelet aggregation 24 hours after loading | 24 hours

SECONDARY OUTCOMES:
Inhibition of platelet aggregation 7 days after loading | 7 days
Inhibition of platelet aggregation 28 days after loading | 28 days
all cause death | 1 year
cardiac death | 1 year
myocardial infarction | 1 year
stent thrombosis (Academic Research Consortium definition) | 1 year
acute hemorrhagic or ischemic stroke excluding transient ischemic attack | 1 year
bleeding complications (Global Use of Strategies to Open Occluded Coronary Arteries [GUSTO] and Thrombolysis In Myocardial Infarction [TIMI] definition) | 1 year
composite of cardiac death, myocardial infarction and stroke | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, Principal Investigator — Professor of Medicine, Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Division of Cardiology, Kyoto University Hospital, Kyoto, Kyoto, Japan